CLINICAL TRIAL: NCT03707119
Title: The Effectiveness of Student 4 Best Evidence as a Tool to Improve Evidence-Based Practice Competencies in Undergraduate Health Professional Students: a Pilot Study
Brief Title: Student 4 Best Evidence as a Tool to Improve Evidence-Based Practice Competencies
Status: Completed | Type: Observational
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Principal Investigator, Chiara Arienti, MSc and PhD(s), Fondazione Don Carlo Gnocchi Onlus
Other Study IDs: S4BE
Record Dates: First submitted 2018-10-08; First posted 2018-10-16 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Undergraduate Health Professional Students
Keywords: educational programme; EBP competencies; training;

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- S4BE: The intervention consisted of the use of Student 4 Best Evidence blog to teach EBP competence. The section S4BE "about" has been used to teach the EBP principles and their key steps and the section S4BE "topics" has been used to teach critical thinking and the clinical practice in rehabilitation for a total of 24 training hours.
  Interventions: Other: Educational programme

INTERVENTIONS:
Other: Educational programme — the health professional students were undergone to Student 4 Best Evidence blog, as a specific educational programme to learn EBP competencies.

SUMMARY:
Objective. The aim of the study was to evaluate the effectiveness of an educational program, based on Students 4 Best Evidence (S4BE) Blog, on Evidence-Based Practice (EBP) competencies (attitudes, knowledge and skills) through an EBP laboratory, in undergraduate students of Physiotherapy.

Design. An observational perspective study. Setting. Physiotherapy School of Italian University. Participants. 70 undergraduate physiotherapist students of the first year, of both genders, were included. Mean age was 20.48+/-3.20 years and 66% were male and 34% were female.

Interventions. The intervention consisted of the use of S4BE to teach EBP competence. The section S4BE "about" has been used to teach the EBP principles and their key steps and the section S4BE "topics" has been used to teach critical thinking and the clinical practice in rehabilitation for a total of 24 training hours.

Main Outcome Measure. The evidence-based practice questionnaire (EBP2Q) has been used to evaluate EBP attitude, knowledge and skills, at the start of laboratory (T0), after 24 training hours (T1) and after 3 months of clinical practice training (follow-up). Statistical analysis was performed with SPSS 17.0 An intra-group analysis has been conducted to verify the improvement during the time. Statistically significant was set at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* undergraduate physiotherapist students of the first year
* both genders

Exclusion Criteria:

* N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 70 undergraduate physiotherapist students of the first year, of both genders, were included. Mean age was 20.48+/-3.20 years, 66% male.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-06-15 (Actual)

PRIMARY OUTCOMES:
Evidence-based practice questionnaire (EBP2Q) | Change from baseline EBP competencies at 24 training hours
  based on 6 domains to evaluate EBP attitude, knowledge and skills

CONTACTS AND LOCATIONS:
Overall Officials: Chiara Arienti, PhD, Principal Investigator — Fondazione Don Carlo Gnocchi
Locations (1):
- Centro "E. Spalenza" - Fondazione Don Carlo Gnocchi, Rovato, Brescia, Italy

IPD SHARING:
Plan to Share IPD: No
IPD are available in the archive of Rehabilitation Centre "E. Spalenza".

REFERENCES:
- [Derived] Arienti C, Lazzarini SG, Pollet J, Negrini S. Students 4 Best Evidence as a digital Problem-Based Learning method to improve Evidence-Based Practice competencies in undergraduate physiotherapy students: an observational study. BMJ Evid Based Med. 2021 Oct;26(5):251-252. doi: 10.1136/bmjebm-2020-111395. Epub 2020 Oct 21. PMID 33087451